CLINICAL TRIAL: NCT02108600
Title: A Phase II Trial of the Efficacy and Safety of Tocilizumab for Treatment of Inflammation in the Renal Allograft
Brief Title: Tocilizumab for Renal Graft Inflammation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Flavio Vincenti (Other)
Responsible Party: Sponsor-Investigator, Flavio Vincenti, Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML29092
Record Dates: First submitted 2014-03-27; First posted 2014-04-09 (Estimated); Results first posted 2021-01-27 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Late Complication From Kidney Transplant
Keywords: Kidney transplantation; Inflammation
MeSH Terms: conditions — Inflammation | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (No Intervention): Will continue usual immunosuppression and not receive any specific intervention.
- Tocilizumab (TCZ) Group (Experimental): Will receive tocilizumab 8 mg/kg intravenously at four-week intervals for a total of 6 doses. In addition, will continue usual immunosuppressive regimen.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Will receive tocilizumab 8 mg/kg intravenously at four-week intervals for a total of 6 doses. In addition, will continue usual immunosuppressive regimen.
  Arms: Tocilizumab (TCZ) Group

SUMMARY:
Randomized open label clinical trial in which 48 renal transplant recipients with inflammation in the 6 month allograft biopsy will either continue usual immunosuppression or receive monthly Actemra (Tocilizumab) infusions for 6 months in addition to usual immunosuppression.

DETAILED DESCRIPTION:
This is a prospective randomized controlled study of kidney transplant recipients with SCI on 6-month surveillance kidney biopsies. SCI for the purpose of this study is defined as 10-50% total parenchymal mononuclear inflammation (Banff ti1-ti2) with <i2,t2 concurrent lesions.

After enrollment, study participants subjects will be randomized to group 1 (standard of care group) or group 2 (tocilizumab (TCZ) group). Block randomization will be performed by the UCSF investigational pharmacy using computer-generated random numbers. The pathologist will be blinded to the randomization.

Group 1 (standard of care group) will continue their usual immunosuppression and not receive any specific intervention.

Group 2 (TCZ group) will receive tocilizumab 8 mg/kg intravenously at four-week intervals for a total of 6 doses.In addition, they will continue their usual immunosuppressive regimen.

As noted above, both groups will continue their usual maintenance immunosuppression regimen. Therefore, recipients who are already receiving prednisone will continue it at 5 mg/day. Recipients on prednisone-free regimens will remain prednisone-free. Mycophenolate mofetil will be continued at the same dose as at the time of the biopsy. Tacrolimus dosing will be adjusted to aim for trough levels of 5-8 mcg/L.

The study period will be 12 months (6 months of therapy plus 6 months of extended follow up- see Study Schema). Any episodes of infections, renal allograft dysfunctions, rejections or other clinical events during the study period will be treated per the usual standard of care.

All participants will be seen by the study PI or co-investigator at monthly study visits. A focused history and physical exam will be performed, including queries for drug toxicities and signs/ symptom of infections. All participants will obtain laboratory tests at intervals of 4 weeks, consisting of a complete blood count, serum electrolytes, BUN and serum creatinine, fasting glucose, liver function tests and 12-hour trough tacrolimus levels. Lipid panels will be obtained at baseline, then every 12 weeks an at study termination.The outpatient electronic medical record will be queried twiceweekly by the study coordinator for any new laboratory results on study participants. Laboratory data on all study participants will be reviewed weekly by the study PI.

The 12-month surveillance biopsy will be performed at the end of therapy (6 months after study enrollment).

ELIGIBILITY:
Inclusion Criteria:

* All kidney transplant recipients with SCI on 6-month surveillance biopsy.
* Maintenance immunosuppression regimens containing tacrolimus and MMF with or without prednisone.
* Ability to provide written informed consent for the study.
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment.

Exclusion Criteria:

General:

• Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization.

Excluded Previous or Concomitant Therapy:

* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of screening.
* Previous treatment with any cell-depleting therapies, including investigational agents or approved therapies, some examples are CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19 and anti-CD20, except Thymoglobulin.
* Treatment with intravenous gamma globulin, plasmapheresis or Prosorba column within 6 months of baseline.
* Immunization with a live/attenuated vaccine within 4 weeks prior to baseline.
* Previous treatment with TCZ (an exception to this criterion may be granted for single dose exposure upon application to the sponsor on a case-by-case basis).
* Any previous treatment with alkylating agents such as chlorambucil, or with total lymphoid irradiation.

Exclusions for General Safety:

* Presence of acute cellular (Banff Type 1-3) or antibody-mediated rejection on 6-month surveillance biopsy or on biopsies for-cause in the previous 6 months.
* History of positive urine or serum screening for BK virus (defined as a quantitative BK virus PCR in urine > 0.5 million copies/ml or any detectable BK viremia) within the first 6 months post-transplant.
* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies.
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (include uncontrolled diabetes mellitus) or gastrointestinal disease (including diverticulitis, ulcerative colitis, or Crohn's disease.)
* Current liver disease as determined by principal investigator unless related to primary disease under investigation.
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, Hepatitis B and C, and herpes zoster, but excluding fungal infections of nail beds).
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening.
* Active TB requiring treatment within the previous 3 years. Patients should be screened for latent TB and, if positive, treated following local practice guidelines prior to initiating TCZ. Patients treated for tuberculosis with no recurrence in 3 years are permitted. (Appendix 8).
* Primary or secondary immunodeficiency (history of or currently active) unless related to primary disease under investigation.
* Evidence of active malignant disease, malignancies diagnosed within the previous 10 years (including hematological malignancies and solid tumors, except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised and cured), or breast cancer diagnosed within the previous 20 years unless related to primary disease under investigation.
* Pregnant women or nursing (breast feeding) mothers.
* Patients with reproductive potential not willing to use an effective method of contraception.
* History of alcohol, drug or chemical abuse within 1 year prior to screening.
* Patients with lack of peripheral venous access.

Laboratory Exclusion criteria (at screening):

* Serum creatinine > 1.6 mg/dL (141 µmol/L) in female patients and > 1.9 mg/dL (168 µmol/L) in male patients. Patients with serum creatinine values exceeding limits may be eligible for the study if their estimated glomerular filtration rates (GFR) are >30 ml/min/1.73 m2.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 times upper limit of normal (ULN)
* Total Bilirubin > 1.5 times ULN
* Platelet count < 100 x 109/L (100,000/mm3)
* Hemoglobin < 85 g/L (8.5 g/dL; 5.3 mmol/L)
* White Blood Cells < 3.0 x 109/L (3000/mm3)
* Absolute Neutrophil Count < 2.0 x 109/L (2000/mm3)
* Absolute Lymphocyte Count < 0.5 x 109/L (500/mm3)
* Positive Hepatitis BsAg, or Hepatitis C antibody

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-12-16 (Actual); Study Completion 2018-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Vincenti, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meier-Kriesche HU, Schold JD, Srinivas TR, Kaplan B. Lack of improvement in renal allograft survival despite a marked decrease in acute rejection rates over the most recent era. Am J Transplant. 2004 Mar;4(3):378-83. doi: 10.1111/j.1600-6143.2004.00332.x. PMID 14961990
- [Background] Nankivell BJ, Fenton-Lee CA, Kuypers DR, Cheung E, Allen RD, O'Connell PJ, Chapman JR. Effect of histological damage on long-term kidney transplant outcome. Transplantation. 2001 Feb 27;71(4):515-23. doi: 10.1097/00007890-200102270-00006. PMID 11258430
- [Background] Nankivell BJ, Borrows RJ, Fung CL, O'Connell PJ, Allen RD, Chapman JR. The natural history of chronic allograft nephropathy. N Engl J Med. 2003 Dec 11;349(24):2326-33. doi: 10.1056/NEJMoa020009. PMID 14668458
- [Background] Cosio FG, Grande JP, Larson TS, Gloor JM, Velosa JA, Textor SC, Griffin MD, Stegall MD. Kidney allograft fibrosis and atrophy early after living donor transplantation. Am J Transplant. 2005 May;5(5):1130-6. doi: 10.1111/j.1600-6143.2005.00811.x. PMID 15816896
- [Result] Chandran S, Leung J, Hu C, Laszik ZG, Tang Q, Vincenti FG. Interleukin-6 blockade with tocilizumab increases Tregs and reduces T effector cytokines in renal graft inflammation: A randomized controlled trial. Am J Transplant. 2021 Jul;21(7):2543-2554. doi: 10.1111/ajt.16459. Epub 2021 Jan 21. PMID 33331082

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Tocilizumab (TCZ) Group
Started | 17 | 16
Completed | 14 | 15 (1 patient lost to follow up after the primary endpoint biopsy)
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: n=17 signed consent but 3 withdrew before primary endpoint (2 of them before visit 1) Therefore n=14 were analyzed for baseline characteristics
Groups:
- Tocilizumab (TCZ) Group: Will receive tocilizumab 8 mg/kg intravenously at four-week intervals for a total of 6 doses. In addition, will continue usual immunosuppressive regimen.
  Tocilizumab: Will receive tocilizumab 8 mg/kg intravenously at four-week intervals for a total of 6 doses. In addition, will continue usual immunosuppressive reg
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Tocilizumab (TCZ) Group | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51.5 [40 to 56] | 53.5 [41.5 to 59] | 52 [40 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 10 | 14 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Inflammation on Renal Allograft Biopsy From Baseline to 6 Months
Description: Proportion of participants in each group who had a 1 point decrease in inflammation based on Banff scoring on renal allograft biopsy at 6 months compared to baseline. The Banff ti- score can be 0, 1, 2 or 3.
Time Frame: Baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Tocilizumab (TCZ) Group
Number analyzed (Participants) | 14 | 16
Participants | 3 | 10
Statistical Analysis 1: Comparison: Standard of Care vs Tocilizumab (TCZ) Group; Test type: Other; p = 0.033, Fisher Exact

2. Secondary Outcome: Change in Urinary Cytokines
Description: Change in urinary cytokines from baseline at 6 months.
Time Frame: Baseline and 6 months
Population: The urine samples were not adequate for analysis and therefore this outcome was not analyzed.
Arm/Group | Standard of Care | Tocilizumab (TCZ) Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Development of Donor Specific Anti-HLA Antibodies
Description: Proportion of participants who developed de novo DSA from baseline to 6 months
Time Frame: From baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Tocilizumab (TCZ) Group
Number analyzed (Participants) | 14 | 16
Participants | 0 | 0

4. Secondary Outcome: Incidence of Acute Rejection
Description: Proportion of patients with acute rejection in each group
Time Frame: In the interval between baseline and 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Tocilizumab (TCZ) Group
Number analyzed (Participants) | 14 | 16
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: used Common Terminology Criteria for Adverse Events (CTCAE) grades
Arm/Group | Standard of Care | Tocilizumab (TCZ) Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 3/16
Other Adverse Events (participants affected / at risk) | 0/14 | 2/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=14) | Tocilizumab (TCZ) Group (N=16)
sepsis (Infections and infestations) | 0 (0) | 1 (1) — pneumonia + sepsis
pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
subcapsular hematoma (Renal and urinary disorders) | 0 (0) | 1 (1) — post primary endpoint biopsy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=14) | Tocilizumab (TCZ) Group (N=16)
pneumonia (Infections and infestations) | 0 (0) | 1 (1)
skin infection (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study could not meet its recruitment target of 48 subjects, and consequently, is underpowered statistically. Additionally, the urine samples were inadequate, leading to inability to perform urine cytokine measurements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT02108600/Prot_SAP_000.pdf